CLINICAL TRIAL: NCT03576976
Title: Improving Accessibility and Personalization of Cognitive Remediation for Schizophrenia
Brief Title: Improving Accessibility and Personalization of CR for Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Alice Medalia, Professor of Medical Psychology in Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7638; 1P50MH115843-01 (NIH)
Record Dates: First submitted 2018-05-25; First posted 2018-07-05 (Actual); Results first posted 2022-02-02 (Actual); Last update posted 2022-07-13 (Actual); Status verified 2022-06

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: Cognitive Remediation
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — Cognitive Remediation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Clinic-based Cognitive Remediation (Active Comparator): Clinic-based cognitive remediation is the current standard of care in NY State outpatient programs. It consists of twice weekly group-based and clinician-led sessions.
  Interventions: Behavioral: Cognitive Remediation
- Hybrid Cognitive Remediation (Experimental): Hybrid cognitive remediation consists of one weekly group-based, clinician-led session plus independent cognitive practice.
  Interventions: Behavioral: Cognitive Remediation

INTERVENTIONS:
Behavioral: Cognitive Remediation — Computer-based exercises targeting impairments in cognitive domains (sensory processing, processing speed, attention, working memory, memory, executive functions) are paired with verbal discussions and group-based activities to strengthen metacognition to and bridge newly learned cognitive skills to everyday life.

SUMMARY:
This project will explore adaptations of treatments for schizophrenia, with the goal of optimizing their effectiveness in real-world clinical settings and readiness for broad deployment. Schizophrenia is associated with cognitive deficits that negatively impact essential areas of daily functioning. NY State Office of Mental Health (OMH) is the first and largest state system of care to implement a statewide program of cognitive remediation (CR), an evidence-based practice for improving cognition and aiding functional recovery. Through Cognitive Remediation to Promote Recovery (CR2PR), CR is now offered in outpatient programs, with plans to expand to more services and further adapt implementation to improve treatment outcomes. This project will work directly with OMH clinics and clinicians to build upon and improve current CR delivery methods. This project will study the impact of two adaptations. One focuses on increasing the accessibility of the program, which participants report is limited by the requirement of twice weekly attendance. This project will compare the feasibility and acceptability of delivering CR in either two clinic-based sessions (Clinic) or one clinic and one remote session (Hybrid) per week. Qualitative interviews will be conducted with stakeholders to explore the impact of the adaptation. The second adaptation is intended to improve personalization of CR by systematically accounting for individual differences in neurocognitive needs. Drawing upon convergent evidence for tailoring CR based on need for early auditory processing (EAP) training, this project examines whether integrating a measure of EAP into the current baseline assessment facilitates personalization of the menu of restorative computer-based exercises used in CR. Feasibility parameters and qualitative/quantitative data analyses of facilitators and barriers to Hybrid CR delivery will together inform further treatment refinement and the design of a larger effectiveness trial of Clinic versus Hybrid CR. This project will examine how EAP assessment is employed by practitioners to personalize the CR treatment plan and examine if EAP improvement is associated with cognitive outcomes in public practice CR settings. Finally cognitive, functional, and service use outcomes in Hybrid versus Clinic CR will be compared.

DETAILED DESCRIPTION:
Cognitive remediation (CR) is an evidence-based practice to treat the pervasive and significant cognitive deficits that contribute to functional decline in schizophrenia. The New York State Office of Mental Health (OMH) has teamed with the Principal Investigator to be the first, and largest state system of care to implement a statewide program of CR tied to recovery programming. Through Cognitive Remediation to Promote Recovery (CR2PR), CR is now offered in outpatient programs throughout the state, with plans to expand to more services and further adapt implementation to improve treatment outcomes. To proceed systematically, this project will work directly with CR2PR programs, guided by practice-based evidence gathered during CR2PR to build upon and improve current CR delivery methods in two ways.

1. Ongoing program evaluation indicates that the burden of attending clinic twice per week for CR limits the number of people who enroll. This project will test the feasibility and collect preliminary data on the effectiveness of personalized CR delivery that involves one clinic visit and one remote session per week. Demonstrating the effectiveness of incorporating remotely delivered CR would double the number of patients who could access the OMH CR program and reduce treatment costs.
2. Current effect sizes for cognition and functional outcomes may remain limited if personalization, mechanisms of action, and relevant targets are not better addressed. Given evidence that early auditory information processing ability (EAP) works as a neurobehavioral marker of need for sensory processing training, this study will test the potential to use baseline EAP assessment to tailor CR, incorporating EAP with other cognitive skills training as clinically indicated. The ultimate goal of integrating scalable assessment practices to personalize CR is to improve recovery outcomes.

The study will use a repeated measures, randomized design. Eligible participants who are referred to CR2PR will complete a routine baseline neurocognitive assessment with the addition of a EAP measure, and will then be randomized to either all-clinic CR (Clinic) or clinic+remote (Hybrid) CR. The Clinic research arm consists of 30 sessions delivered twice weekly in a group format of up to 8 participants with rolling admission. The Hybrid condition consists of 15 clinic sessions in the above format, and independent homework on cognitive exercises for 60 minutes per week for 15 weeks using a laptop, PC or tablet available to them. All clinic sessions consist of 45 minutes of working on 3-4 computerized exercises selected by a clinician from a menu of web-based programs to improve the cognitive functions identified as impaired on the assessment. Computer exercises are followed by 15 minute manualized discussion groups based on the concept of "Bridging".

All participants will complete a treatment satisfaction survey and will be re-tested on outcome measures approximately 1 week following end of treatment. Additional data on the feasibility and acceptability of the Hybrid approach will be gathered through a qualitative interview with participants at treatment endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Referred for participation in Cognitive Remediation to Promote Recovery by outpatient clinic teams
* A primary DSM-5 diagnosis of schizophrenia or schizoaffective disorder
* Verbal IQ estimate of 70 or above
* Stabilized on any psychotropic medication
* English-speaking

Exclusion Criteria:

* Unremitted substance dependence
* Neurological illness affecting brain functioning
* Traumatic brain injury within 2 years
* Auditory or visual impairment (uncorrected)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-07-16 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2022-05-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alice Medalia, PhD, Principal Investigator — New York State Psychiatric Institute
Locations (7):
- United States (7):
  - Williamsburg Clinic, Brooklyn, New York
  - Heights Hill Clinic, Brooklyn, New York
  - Mapleton Mental Health Services, Brooklyn, New York
  - Manhattan Psychiatric Center 125th St Outpatient Clinic, New York, New York
  - Inwood Clinic, New York, New York
  - Rockland Psychiatric Center, Orangeburg, New York
  - Creedmoor Psychiatric Center, Queens Village, New York

IPD SHARING:
Plan to Share IPD: Yes
Raw data will be made available for research to investigators working under a Federal Wide Assurance who meet security measures and data use agreement criteria associated with public repositories including the National Database for Clinical Trials related to Mental Illness (NDCT) and the NIMH Database of Cognitive Training and Remediation Studies (DoCTRS). Data will include baseline demographic data, and baseline and post raw data derived from cognitive, quality of life, functioning and symptom measures.
Time Frame: A list of all data expected to be collected in the project will be submitted within 6 months of award. Subsequently, descriptive and raw data will be submitted on a semi-annual basis. Unpublished de-identified data will be submitted prior to study completion and will be shared within one year after project completion, or when the data are published, whichever is earlier.
Access Criteria: Data in NIH repositories may be accessed through the NIH Data Access Committee which reviews data access and submission requests.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Enrolled participants were screened and assessed on outcome measures prior to randomization. Those who did not complete baseline assessments due to lost contact or no longer meeting inclusion criteria were not assigned to a treatment condition and were exited from the study.
Period: Overall Study
Arm/Group | Clinic-based Cognitive Remediation | Hybrid Cognitive Remediation
Started | 27 | 28
Completed | 18 | 17
Not Completed | 9 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clinic-based Cognitive Remediation | Hybrid Cognitive Remediation | Total
Number analyzed (Participants) | 27 | 28 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.32 (12.73) | 48.99 (12.05) | 45.71 (12.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 20 | 19 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 8 | 17
  Not Hispanic or Latino | 18 | 20 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 14 | 32
  White | 7 | 11 | 18
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 1
IQ Estimate [Mean (Standard Deviation); unit: units on a scale] — The Wechsler Test of Adult Reading (WTAR) yields an age-adjusted standard score which is used as an IQ estimate. The IQ estimate has a mean of 100 and standard deviation of 15. Higher scores indicate higher IQ (estimated intellectual ability).
  units on a scale | 92.67 (10.32) | 90.86 (10.82) | 91.75 (10.52)

OUTCOME MEASURES:

1. Primary Outcome: Treatment Satisfaction
Description: Treatment satisfaction will be measured using a self-report Likert-type rating scale questionnaire reflecting the specific components of the treatments used for this study. The outcome measure will be an average of the scale items, ranging from 1 to 6, with 1 reflecting strong dissatisfaction with the treatment and 6 reflecting strong satisfaction with the treatment.
Time Frame: Through study completion, 15 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Clinic-based Cognitive Remediation | Hybrid Cognitive Remediation
Number analyzed (Participants) | 18 | 17
score on a scale | 5.25 (0.97) | 5.32 (0.98)

2. Secondary Outcome: Change From Baseline in Neurocognition
Description: Neurocognition will be measured with subtests from the Brief Assessment of Cognition in Schizophrenia (BACS): Verbal Memory (verbal memory and learning), Digit Sequencing (working memory), Symbol Coding (speed of processing), and Tower of London (executive function) and the Continuous Performance Test - Identical Pairs (CPT-IP; attention/vigilance). A T score for each subtest is obtained where the population mean is 50 and the standard deviation is 10. For all subtests higher scores indicate better outcome. An average T score is generated to capture neurocognition at each assessment time point. The secondary outcome measure is change in the average T score from baseline to post-treatment.
Time Frame: Baseline and 15 weeks
Population: The analysis population includes all participants who completed the intervention phase who were able to attend a post-treatment assessment.
Measure: Mean (Standard Deviation); unit: T Score
Arm/Group | Clinic-based Cognitive Remediation | Hybrid Cognitive Remediation
Number analyzed (Participants) | 17 | 15
T Score | -1.49 (3.6) | 0.97 (6.56)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for each individual from baseline to post-treatment, approximately 15 weeks.
Arm/Group | Clinic-based Cognitive Remediation | Hybrid Cognitive Remediation
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 0/27 | 0/28

LIMITATIONS AND CAVEATS:
COVID-19 pandemic limited post-treatment data collection at the conclusion of the trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-05-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT03576976/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-24): https://cdn.clinicaltrials.gov/large-docs/76/NCT03576976/SAP_001.pdf